CLINICAL TRIAL: NCT02839083
Title: Thoracic Paravertebral Block Versus Pecs II Block for Perioperative Analgesia in Modified Radical Mastectomy
Brief Title: Pecs II Block as Alternative for Paravertebral Block in Modified Radical Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD ∕ 153
Record Dates: First submitted 2016-07-16; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Modified Radical Mastectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracic Paravertebral group (Placebo Comparator): Ultrasound guided thoracic paravertebral block
  Interventions: Other: Thoracic Paravertebral group
- Pecs II group (Active Comparator): Ultrasound guided Pecs II block
  Interventions: Other: Pecs II group

INTERVENTIONS:
Other: Thoracic Paravertebral group — Thoracic paravertebral block is performed using bupivacaine 0.25% in a total volume of 30 ml
  Arms: Thoracic Paravertebral group
Other: Pecs II group — Ultrasound guided ipsilateral Pecs II block is performed using bupivacaine 0.25% in a total volume of 30 ml
  Arms: Pecs II group

SUMMARY:
Breast surgeries are usually associated with significant postoperative pain. Suitability of analgesic technique after breast surgery is always questionable. The aim of this study is to compare US guided Pecs II block versus thoracic paravertebral block performed by US guidance as regards to potential complications and analgesic efficacy of both techniques in the first 24 h after modified radical mastectomy.

DETAILED DESCRIPTION:
Various modalities have been used for perioperative pain management in relevance to breast surgery. Thoracic epidural and paravertebral blocks (PVB) became the gold standard techniques to achieve this goal. However, both techniques may be associated with devastating complications such as spinal cord injury, total spinal anesthesia, inadvertent intravascular injection and pneumothorax.

On the other hand, the advancement of ultrasound (US) technology and our ability to visualize the pleura and other structures in and around the paravertebral space has increased interest in performing thoracic paravertebral blocks guided by US.

"Pecs" block is a less invasive procedure involving US guided interfascial injections has been suggested as potential alternative analgesic technique. The Pecs I block was initially described by Blanco for minor breast surgery. A year later, on 2012, he described a Pecs II block or "modified Pecs block" for breast surgery involving the axilla.

The Pecs I block targets the medial pectoral nerve (MPN) from C8 and T1 and the lateral pectoral nerve (LPN) from C5, C6, and C7. These nerves arise from the medial and lateral cords of the brachial plexus, respectively, and innervate the pectoralis muscles.

The Pecs II block targets the T2-6 intercostal nerves, the long thoracic nerve which supplies the serratus anterior, and the thoracodorsal nerve which supplies the latissimus dorsi. Potential complications include accidental intravascular injection and pneumothorax.

The easily identifiable landmarks allow this block to provide a simple alternative to paravertebral and neuraxial blocks for breast surgery. The block produces excellent analgesia and can be used as a rescue block in cases with patchy or ineffective paravertebral or epidural block.

ELIGIBILITY:
Inclusion Criteria:

* American Association for Anesthesiologists physical status I or II
* Body mass index > 40 kg/m2

Exclusion Criteria:

* Patient refusal
* Severe or uncompensated cardiovascular disease.
* Significant renal disease.
* Significant hepatic disease.
* Significant endocrinal disease.
* Pregnancy.
* Postpartum period.
* Lactating females.
* Allergy to any of the study medication.
* Coagulation disorders.
* Infection at the site of needle insertion.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain scores | For 24 hours after surgery
  Pain visual analog scale is used to assess the severity of postoperative pain

SECONDARY OUTCOMES:
Duration of postoperative analgesia | for 12 hours after surgery
  period from completion of the block to time of administration of the first rescue analgesic for 12 hour after performing the block
Cumulative postoperative meperidine consumption | for 48 hours after surgery
  Cumulative consumption of rescue meperidine analgesic for 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elaziz Metawa, MD, Study Chair — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt
Locations (1):
- Mansoura university, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided